CLINICAL TRIAL: NCT04375670
Title: COVID19-FOIE National Observatory. An Ambispective Cohort Study of All Consecutive Patients
Brief Title: COVID19-FOIE National Observatory
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association Française pour l'Etude du Foie (AFEF) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00006477
Record Dates: First submitted 2020-04-28; First posted 2020-05-05 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Liver Diseases; COVID19
Keywords: Mortality; Fibrosis; Hepatocellular Carcinoma
MeSH Terms: conditions — Liver Diseases; COVID-19; Fibrosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

The COVID19 and liver relationships are very rare. The preliminary Chinese data indicate that 2-11% of patients treated for COVID19 had an underlying chronic liver disease. However, there is no clinical data on morbi-mortality in this context.

Objectives:

Primary Objective:

Evaluate the mortality related to Covid-19 in patients with a chronic liver disease

Secondary objectives:

* Evaluate the mortality (liver-related and no liver-related) due to the Covid-19 according to the cirrhotic status, an history of hepatocellular carcinoma, an immunosuppressive treatment and its type, the etiology-ies of liver disease at the diagnosis of Covid-19 (viral hepatitis -B and/or C-, liver disease related to alcohol consumption, metabolic syndrome, hemochromatosis, immune liver disease, other or unknown), and comorbidities
* Evaluate the liver morbidity related to Covid-19, including
* incidence of liver biochemical abnormalities in patients with normal liver enzymes values or of a 2-fold increase of usual values for AST, ALT, GGT, Alcalines Phosphatasis
* incidence of liver complications (acute hepatitis, liver insufficiency, decompensation of cirrhosis, encephalopathy, renal insufficiency)

Patients:

All patients with a liver disease (chronic or acute) with a positive diagnosis of Covid-19 assessed either by positive PCR or specific thoracic abnormalities at TDM

Methodology:

Observational ambispective study consisting exclusively of a collection of data from patients with liver diseases and managed for COVID 19 The data is collected and transcribed on a secure electronic eCRF hosted at the Assitance Publique des Hôpitaux de Paris and accessible online from the AFEF website

Duration and organisation of the research:

After information of the patients and making available a non-opposition form, the main demographic and clinical data related to the liver disease and to the COVID19 already collected in the patient's medical record will be collected in a dedicated e-CRF.

Effective of the study:

All consecutive patients included in the study whose data are collected e-CRF until 31/12/2020.

DETAILED DESCRIPTION:
1. Background and objectives:

   Coronavirus infection 2019 (COVID-19), linked to the SARS-Cov-2 virus, is rapidly spreading worldwide. After the city of Wuhan and the province of Hubei, European healthcare systems are facing an outbreak of seriously ill patients, but few are fully equipped to manage this health crisis.

   On the occasion of this pandemic, the hepatologist associations of United States , Europe and France as well as the French Federation of Digestive Cancer have proposed modalities for the management of patients with chronic liver disease likely to guarantee them maximum safety. The level of scientific evidence for these proposals is very low, given the small amount of objective clinical data available to date on the relationship between COVID-19 and liver.

   Some preliminary Chinese data indicates that:
   * 2-11% of patients treated for COVID19 had underlying chronic liver disease
   * an increase in transaminases is observed in 25-35% of patients, generally moderate (median 23-39 IU/L), with a higher rate in symptomatic and/or severe forms and/or requiring hospitalization in intensive care unit as well as in patients who later die . The mechanism involved is uncertain to date. Indeed, the data suggesting the possibility of localization of the virus in the liver are too preliminary, and it is reasonable to incriminate the elements of inflammatory reaction syndrome. Liver damage can be explained during these infections by hepatic hypoxia, related to a frequent viral myocarditis in this situation. Finally, other more classic causes may also be associated, including drug (paracetamol, antibiotics), or an exacerbation of an underlying chronic liver disease, known or unknown. Control of viral serologies B and C is therefore recommended in this situation.
   * elderly patients, patients with cirrhosis, patients with immune hepatitis under immunosuppressive drugs and patients before and after transplantation under immunosuppressive therapy would be the subjects most at risk of severe COVID19
   * very strict preventive measures have proven their effectiveness in terms of mortality in 111 patients with decompensated cirrhosis, including 2/3 hospitalized and 1/3 ambulatory.

   In this totally new and unexpected context, the board meeting of the AFEF proposes the national observatory COVID19-FOIE, intended to collect data of patients with liver disease (all stages combined) or liver transplants that developed COVID19 confirmed by PCR on nasopharyngeal sampling and/or thoracic CT.
2. Population:

   All patients with acute or chronic liver disease treated by a member of the AFEF with an established diagnosis of COVID 19 confirmed by PCR on nasopharyngeal and/or thoracic CT.
3. Methodology:

   This is an epidemiological, observational, prospective, descriptive, prognostic and evaluative observational cohort study. This study does not change the patient's management; it consists of analyzing clinical-biological data collected as part of the patient's usual follow-up.
4. Objectives:

   Primary Objective:

   Evaluate the mortality related to Covid-19 in patients with a chronic liver disease

   Secondary objectives:
   * Evaluate the mortality (liver-related and no liver-related) due to the Covid-19 according to the cirrhotic status, an history of hepatocellular carcinoma, an immunosuppressive treatment and this type, the etiology-ies of liver disease at the infection (viral hepatitis -B and/or C-, related to alcohol consumption, metabolic syndrome, hemochromatosis, immune liver disease, other or unknown), and comorbidities
   * Evaluate the liver morbidity related to Covid-19, including :
   * incidence of liver biochemical abnormalities in patients with normal liver enzymes values or of a 2-fold increase of usual values for AST, ALT, GGT, alcalines phosphatasis
   * incidence of liver complications (acute hepatitis, liver insufficiency, decompensation of cirrhosis, encephalopathy, renal insufficiency)
5. Criteria:

   Primary criteria: mortality rate related to Covid-19 in patients with a chronic liver disease

   Secondary criteria:
   * mortality rate according the stage of fibrosis and the cirrhotic status defined with liver biopsy or non invasive tests of fibrosis or according the opinion of clinician
   * mortality related to Covid-19 according an history of hepatocellular carcinoma, an immunosuppressive treatment and this type (treatment related to a liver transplantation or to an auto-immune liver disease or to other indication), the etiology-ies of liver disease at the infection (viral hepatitis -B and/or C-, related to alcohol consumption, metabolic syndrome, hemochromatosis, immune liver disease, other or unknown), and comorbidities, particularly diabetes, hypertension, overweight -BMI from 26 to 30- or obesity-BMI > 30)
   * Incidence of liver complications (acute hepatitis, liver insufficiency, decompensation of cirrhosis, encephalopathy, renal insufficiency)
6. Effective and duration of the study:

   All consecutive patients included in the observatory with registered data in the eCRF until 31/12/20.
7. Population of the study:

   * Inclusion criteria:
   * all patients with acute or chronic liver disease managed by a member of AFEF with positive diagnosis of COVID-19 by PCR and/or specific abnormalities at the thoracic TDM
   * patients with history of liver transplantation
   * patients affiliated with social security
   * Non inclusion criteria: age equal or higher 18 years
8. Conduct of the research:

After informing patients and making available a non opposition form, the main demographic and clinical data related to a chronic liver disease, in one hand and, on the other hand, the COVID19, already collected in the patient's medical record will be collected in a dedicated eCRF. All contributors will be associated with the publications resulting from this observatory and the COVID-Foie working group.

ELIGIBILITY:
Inclusion Criteria:

* All patients with acute or chronic liver disease managed by a member of AFEF with positive diagnosis of COVID-19 by PCR and/or specific abnormalities at the thoracic TDM
* Patients with history of liver transplantation
* Patients affiliated with social security

Exclusion Criteria:

* Age inferior to 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a liver disease (chronic or acute) with a positive diagnosis of Covid-19 assessed either by positive PCR or specific thoracic abnormalities at TDM
Sampling Method: Non-Probability Sample
Enrollment: 1132 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Mortality rate related to Covid-19 in patients with a chronic liver disease | Up to 30 days

SECONDARY OUTCOMES:
mortality rate according the stage of fibrosis and the cirrhotic status | Up to 30 days
  defined with liver biopsy or non invasive tests of fibrosis or according the opinion of clinician
mortality related to Covid-19 according an history of hepatocellular carcinoma, an immunosuppressive treatment and this type the etiology-ies of liver disease at the infection and comorbidities. | Up to 30 days
Incidence of liver complications | through patient follow-up, an average of 1 year
  acute hepatitis, liver insufficiency, decompensation of cirrhosis, encephalopathy, renal insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Ganne-Carrié, MD-PhD, Principal Investigator — AP-HP, Jean Verdier Hospital
Locations (1):
- Ganne, Bondy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Clinical Insights for Hepatology and Liver Transplant Providers During the COVID-19 Pandemic.https://www.aasld.org/sites/default/files/2020-03/AASLD-COVID19-ClinicalInsights-3.23.2020-FINAL-v2.pdf
- [Background] Boettler T, Newsome PN, Mondelli MU, Maticic M, Cordero E, Cornberg M, Berg T. Care of patients with liver disease during the COVID-19 pandemic: EASL-ESCMID position paper. JHEP Rep. 2020 Jun;2(3):100113. doi: 10.1016/j.jhepr.2020.100113. Epub 2020 Apr 2. PMID 32289115
- [Background] Di Fiore F, Bouche O, Lepage C, Sefrioui D, Gangloff A, Schwarz L, Tuech JJ, Aparicio T, Lecomte T, Boulagnon-Rombi C, Lievre A, Manfredi S, Phelip JM, Michel P; Thesaurus National de Cancerologie Digestive (TNCD); Societe Nationale Francaise de Gastroenterologie (SNFGE); Federation Francophone de Cancerologie Digestive (FFCD); Groupe Cooperateur multidisciplinaire en Oncologie (GERCOR); Federation Nationale des Centres de Lutte Contre le Cancer (UNICANCER); Societe Francaise de Chirurgie Digestive (SFCD); Societe Francaise d'Endoscopie Digestive (SFED); Societe Francaise de Radiotherapie Oncologique (SFRO) and Societe Francaise de Radiologie (SFR); Association Chirurgie Hepato-Biliaire et Transplantation (ACHBT). COVID-19 epidemic: Proposed alternatives in the management of digestive cancers: A French intergroup clinical point of view (SNFGE, FFCD, GERCOR, UNICANCER, SFCD, SFED, SFRO, SFR). Dig Liver Dis. 2020 Jun;52(6):597-603. doi: 10.1016/j.dld.2020.03.031. Epub 2020 May 14. PMID 32418773
- [Background] Zhang C, Shi L, Wang FS. Liver injury in COVID-19: management and challenges. Lancet Gastroenterol Hepatol. 2020 May;5(5):428-430. doi: 10.1016/S2468-1253(20)30057-1. Epub 2020 Mar 4. No abstract available. PMID 32145190
- [Background] Xu L, Liu J, Lu M, Yang D, Zheng X. Liver injury during highly pathogenic human coronavirus infections. Liver Int. 2020 May;40(5):998-1004. doi: 10.1111/liv.14435. Epub 2020 Mar 30. PMID 32170806
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Xiao Y, Pan H, She Q, Wang F, Chen M. Prevention of SARS-CoV-2 infection in patients with decompensated cirrhosis. Lancet Gastroenterol Hepatol. 2020 Jun;5(6):528-529. doi: 10.1016/S2468-1253(20)30080-7. Epub 2020 Mar 17. No abstract available. PMID 32197093